CLINICAL TRIAL: NCT00957424
Title: International Study of the Acceptability of Less Harmful Alternatives to Cigarettes (ISALHAC) - A Pilot Study
Brief Title: Acceptability of Less Harmful Alternatives to Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CDR0000648665; P30CA016056 (NIH); RPCI-I-118207
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Bladder Cancer; Cervical Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Kidney Cancer; Leukemia; Liver Cancer; Lung Cancer; Pancreatic Cancer; Tobacco Use Disorder
Keywords: tobacco use disorder; bladder cancer; cervical cancer; esophageal cancer; gastric cancer; renal cell carcinoma; adult primary liver cancer; non-small cell lung cancer; small cell lung cancer; pancreatic cancer; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; adult acute myeloid leukemia
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Tobacco Use Disorder; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Leukemia, Myeloid, Acute | interventions — Nicotine Replacement Therapy

ARMS (1):
- Overall (Other): Single-armed study
  Interventions: Behavioral: telephone-based intervention; Drug: nicotine replacement therapy; Other: informational intervention; Other: internet-based intervention; Other: questionnaire administration

INTERVENTIONS:
Behavioral: telephone-based intervention — 10-15 minute web-based survey on a computer
Drug: nicotine replacement therapy — One week supply
Other: informational intervention
Other: internet-based intervention
Other: questionnaire administration — Given out week 2, 3 and 4.

SUMMARY:
RATIONALE: A study that evaluates participants' beliefs about smokeless tobacco products and nicotine replacement therapy may be useful in helping smokers stop smoking.

PURPOSE: This clinical trial is studying the acceptability of less harmful alternatives to cigarettes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the impact of factual information (a fact sheet) about the relative harms of smokeless (SL)/nicotine replacement (NR) products on participants' beliefs about relative harmfulness.
* To assess the impact of trying samples of NR and/or SL products on intentions to use such products as alternatives to cigarettes.

Secondary

* To explore the effects of factual information in regard to smoked tobacco on smokers' intentions to use such products as alternatives to cigarettes.
* To assess potential barriers to use of both NR and SL products as substitutes for cigarettes.
* To obtain estimates of possible effect sizes for powering a proposed comprehensive test of the likely outcomes of using these products in preference to cigarettes (and other smoked products).

OUTLINE:

Participants undergo a 10-15 minute web-based survey on a computer in the Tobacco Research Laboratory to assess basic demographic information; beliefs about the relative harmfulness of nicotine replacement (NR) and smokeless (SL) products, including use of relevant questions from the International Tobacco Control (ITC) 4 country survey; past experiences with NR and SL products and perceptions about them; and willingness to try samples of NR/SL products they have not previously used, or, if not willing, reasons for refusal. Participants also receive an information sheet while simultaneously hearing an audio recording of it.

Participants complete questionnaires at 2, 3, and 4 weeks.

Beginning 2 weeks after study intervention, some participants receive a day's supply of ≤ 4 smokeless tobacco or nicotine products and periodically undergo a breath CO and saliva and buccal cell sample collection. Surveys are completed and samples collected at 3 and 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently smokes ≥ 10 cigarettes per day
* Not planning to quit smoking in the next 30 days and has not tried to quit in the past 30 days
* Medically eligible to receive nicotine-replacement products, based on the NYS Smokers Quitline eligibility criteria

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Able to read and speak English
* In good general health
* No history of heart attack or stroke in the past 2 weeks
* No history of chest pains in the past month
* No report of physician-diagnosed arrhythmia/irregular heartbeat or use of pacemaker
* No report of physician-diagnosed heart disease/coronary artery disease, uncontrolled hypertension, stomach ulcer, diabetes, depression, or asthma

PRIOR CONCURRENT THERAPY:

* No other concurrent tobacco products or nicotine medications
* No concurrent Zyban, Bupropion, Wellbutrin, Chantix, or other smoking cessation medication

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mahoney, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Noncombusted Nicotine Product With Informational Intervention: Single-armed study
Period: Overall Study
Arm/Group | Noncombusted Nicotine Product With Informational Intervention
Started | 67
Follow-up #1 | 59
Follow-up #2 | 50
Completed | 44
Not Completed | 23
Not completed — Lost to Follow-up | 19
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Current smokers, aged 18+, smoke at least 10 cigarettes per day, not planning to quit smoking in the next 30 days
Arm/Group | Overall
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (9.59)
Gender [Count of Participants; unit: Participants]
  Female | 35
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 42
  More than one race | 5
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Interest in Trial of Harm-reduction Products (HRPs)
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 67
participants | 7

2. Primary Outcome: Number of Participants Willing to Try HRPs
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 67
participants | 60

3. Primary Outcome: Number of Participants That Completed 1-week Trial
Time Frame: One week
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 67
participants | 50

4. Primary Outcome: Number of Participants Willing to Continue With Preferred HRP
Time Frame: 1 week follow up
Population: Those who completed one-week multiple product sampling
Measure: Number; unit: participants
Arm/Group | Overall
Number analyzed (Participants) | 50
participants | 49

ADVERSE EVENTS:
Time Frame: Collected over 2 weeks while participants were using tobacco products
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

LIMITATIONS AND CAVEATS:
About 1/3 of initial participants did not complete this study. The limited number of participants precludes identifying demographic predictors of willingness or patterns of substitution. Single armed study lacks comparison group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No